CLINICAL TRIAL: NCT05432804
Title: A Phase 1 and Randomized Phase 2 Trial of Selinexor and Temozolomide in Recurrent Glioblastoma
Brief Title: Testing the Addition of an Anti-cancer Drug, Selinexor, to the Usual Chemotherapy Treatment (Temozolomide) for Brain Tumors That Have Returned After Previous Treatment
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Other - Protocol amendment to use placebo
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-05066; NCI-2022-05066 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-222; 10505 (Other: City of Hope Comprehensive Cancer Center LAO); 10505 (Other: CTEP); UM1CA186717 (NIH)
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: MGMT-Methylated Glioblastoma; Recurrent Glioblastoma, IDH-Wildtype; Recurrent MGMT-Methylated Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; selinexor; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (temozolomide) (Active Comparator): Patients receive temozolomide PO on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo MRI throughout the study and blood sample collection while on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Drug: Temozolomide
- Group II (temozolomide, selinexor) (Experimental): Patients receive temozolomide PO on days 1-5 of each cycle and selinexor PO on days 8 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo MRI throughout the study and blood sample collection while on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Drug: Selinexor; Drug: Temozolomide

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Selinexor — Given PO
  Other Names: ATG-010; CRM1 Nuclear Export Inhibitor KPT-330; KPT 330; KPT-330; KPT330; Nexpovio; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330; Xpovio
  Arms: Group II (temozolomide, selinexor)
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase I/II trial tests the safety, side effects and best dose of selinexor given in combination with the usual chemotherapy (temozolomide) and compares the effect of this combination therapy vs. the usual chemotherapy alone (temozolomide) in treating patients with glioblastoma that has come back (recurrent). Selinexor is in a class of medications called selective inhibitors of nuclear export (SINE). It works by blocking a protein called CRM1, which may keep cancer cells from growing and may kill them. Temozolomide is in a class of medications called alkylating agents. It works by damaging the cell's DNA and may kill tumor cells and slow down or stop tumor growth. Giving selinexor in combination with usual chemotherapy (temozolomide) may shrink or stabilize the tumor better than the usual chemotherapy with temozolomide alone in patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of temozolomide followed by selinexor in recurrent glioblastoma patients as determined by dose-limiting toxicities (DLTs) and the total toxicity profile. (Phase I) II. To evaluate the efficacy of sequentially administering temozolomide and selinexor in recurrent glioblastoma as determined by progression-free survival (PFS). (Phase 2)

SECONDARY OBJECTIVES:

I. To evaluate overall response rate as determined by Response Assessment in Neuro-Oncology (RANO) response criteria.

II. To evaluate the efficacy of sequentially administering temozolomide and selinexor in recurrent glioblastoma as determined by 6-month PFS (6mPFS) and overall survival (OS).

III. To validate signatures of vulnerability to predict response to selinexor through ribonucleic acid (RNA) sequencing for 6 top-scoring gene pairs, whole exome sequencing, P53, EGFR, and Mcl-1.

OUTLINE: This is a phase I, dose-escalation study of selinexor in combination with fixed dose temozolomide followed by a phase II study that compares selinexor temozolomide combination therapy vs. temozolomide monotherapy. Patients are randomized to 1 of 2 groups for the phase II part of this trial.

GROUP I (Phase II): Patients receive temozolomide orally (PO) on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

GROUP II (Phase I and II): Patients receive temozolomide PO on days 1-5 of each cycle and selinexor PO on days 8 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. (Phase I completed as of April 2024)

Patients undergo magnetic resonance imaging (MRI) throughout the study and blood sample collection while on study.

After completion of study treatment, patients are followed up every 2 months up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed glioblastoma (IDH wild-type, MGMT promoter methylated) that has undergone resection or biopsy upon first recurrence. Recurrence at site of prior involvement is defined by histopathological evidence of viable neoplastic cells associated with any of the following: mitotic activity, increased proliferation rate, micro-endothelial proliferation, or pseudo-palisading necrosis
* Prior to resection or biopsy, patients must have measurable disease, defined as at least one bi-dimensional contrast-enhancing lesion with clearly defined margins, with 2 perpendicular diameters of at least 10 mm, visible on >= 2 axial slices
* Patients must have received first-line treatment of temozolomide plus radiotherapy
* Patients must not have received any prior therapy aside from resection or biopsy for their recurrent disease
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of selinexor (KPT-330) in combination with temozolomide in patients < 18 years of age, children are excluded from this study
* Karnofsky performance status >= 60% (Eastern Cooperative Oncology Group [ECOG] =< 2)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 10 g/dL
* Total bilirubin =< 2 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/ alanine transaminase (ALT) serum glutamic-pyruvic transaminase (SGPT) =< 3 x institutional ULN
* Glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retro-viral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* The effects of selinexor (KPT-330) and temozolomide on the developing human fetus are unknown. For this reason and because selective nuclear export inhibitors as well as deoxyribonucleic acid (DNA) alkylating agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for 180 days after the last dose of temozolomide. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 90 days after completion of study treatment administration
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients who have had chemotherapy must have full recovery of organ and marrow function following the nadir of the last chemotherapy cycle
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* Patients who have previously received bevacizumab
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to selinexor (KPT-330) or temozolomide
* History of hypersensitivity to dacarbazine (DTIC), since both dacarbazine and temozolomide are metabolized to 5-(3-methyltriazen-1-yl)-imidazole-4-carboxamide (MTIC)
* Patients with uncontrolled intercurrent illness
* Pregnant women are excluded from this study because selinexor (KPT-330) is a selective inhibitor of nuclear export with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with selinexor (KPT-330), breastfeeding is not allowed for mothers during treatment with selinexor (KPT-330) and for 7 days after the last dose. These potential risks may also apply to other agents used in this study
* Hospitalized patients with severe coronavirus disease of 2019 (COVID-19) who are >= 75 years old, or with a high-risk COVID-GRAM score, or with lactate dehydrogenase (LDH) > 370 (U/L) AND D-Dimer > 600 mcg/L FEU should not receive low-dose selinexor (KPT-330) pending additional results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) (Phase I) | Up to 28 days
  Any eligible patient who receives at least one dose of protocol-defined therapy will be considered evaluable for dose-limiting toxicity (DLT) if either of the following occurs: (1) the patient experiences a DLT during cycle 1 of therapy; or (2) the patient receives at least 4 doses of temozolomide and 1 dose of selinexor. All other patients enrolled during the phase 1 portion of the study will be considered inevaluable for DLT and may be replaced for the purposes of establishing the RP2D.
Progression-free survival (PFS) (Phase II) | From randomization to date of disease progression (either progression of existing lesions or appearance of new lesions), death, or date of last contact, whichever occurs first, assessed up to 3 years
  Patients who experience disease progression or death will be considered to have experienced a PFS-event; otherwise the patient is considered censored at last contact.

SECONDARY OUTCOMES:
Response according to response assessment in neuro-oncology criteria (RANO) criteria | Up to 3 years
  A patient who is evaluated as complete response (CR), partial response (PR), or stable disease (SD) will be considered a RANO-responder. All other patients will be considered RANO-non-responders. Response rate will be calculated and comparisons made using categorical data methods.
Six-month progression-free survival (PFS-6) | At 6 months
  Any patient considered evaluable for RANO response will be considered evaluable for PFS-6. Any evaluable patient who is considered progression free for the primary analysis will be considered a PFS-6 responder. All other evaluable patients will be considered PFS-6 non-responders.
Median overall survival | Time between the date of randomization and the date of death or date of last contact, whichever occurs first, assessed up to 3 years
  Will be calculated from the Kaplan-Meier estimate of the probability of death as a function of time since enrollment. Ninety-five percent (95%) confidence intervals will be calculated as well.
Molecular signatures of vulnerability | Up to 3 years
  Will be assessed using logistic regression for the outcome measure (RANO response) and using proportional hazard regression with the biological characteristic of interest as the predictor variable for risk for PFS event. Patients considered evaluable for RANO response and PFS, respectively, will contribute to the analyses for these exploratory outcomes. Two-sided statistical testing will be employed, and a p-value of 0.05 or less will be considered as indicating significant evidence of association between the particular signature and the outcome of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Frances E Chow, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (36):
- United States (36):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm